CLINICAL TRIAL: NCT03165058
Title: Assessment of Colonic Epithelial Integrity With Mucosal Impedance
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Yash Amit Choksi, Principal Investigator, Vanderbilt University Medical Center
Other Study IDs: 160534
Record Dates: First submitted 2017-05-22; First posted 2017-05-24 (Actual); Results first posted 2020-06-05 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inflammatory Bowel Disease: Patients undergoing standard of care colonoscopy for inflammatory bowel disease (IBD) surveillance will have a MI catheter sensor positioned along the mucosal wall to measure resistance across the mucosa.
  Interventions: Diagnostic Test: mucosal impedance (MI) testing
- control: Patients undergoing standard of care colonoscopy for age appropriate screening will have a MI catheter sensor positioned along the mucosal wall to measure resistance across the mucosa.
  Interventions: Diagnostic Test: mucosal impedance (MI) testing

INTERVENTIONS:
Diagnostic Test: mucosal impedance (MI) testing — During routine colonoscopy, consented study participants will have a MI catheter sensor positioned along the mucosal wall to measure resistance across the mucosa. The physician will take measurements in each segment of the colon, including segments that appear inflamed and normal adjacent areas (up to 10 locations). To obtain a stable reading, the sensor must remain in contact with the mucosa for five seconds. The study procedure will add approximately 1-2 minutes of anesthesia time for each participant. Basic demographic information, prior IBD treatments, and prior colonoscopic data will be collected from the medical record following the procedure for those patients who consent to research.

SUMMARY:
In this study, the investigators propose to use mucosal impedance (MI), a minimally invasive technology, to detect mucosal damage (i.e. barrier dysfunction) based on mucosal conductivity changes in the colonic epithelium.

DETAILED DESCRIPTION:
The intestinal epithelium functions to separate luminal contents from the interstitium. Increased intestinal permeability can represent compromise of the epithelium's integrity. Prior research has demonstrated that defects in intestinal barrier function are associated with inflammatory bowel disease (IBD) and increased intestinal permeability can be important in the maintenance of remission in IBD patients. There is currently not a convenient way to measure colonic epithelial barrier function in real time which could provide clinically relevant information .

ELIGIBILITY:
Inclusion Criteria:

* Men and women over the age of 18 with a diagnosis of IBD (Ulcerative Colitis or Crohn's Disease)
* Men and women undergoing screening colonoscopy (typical age would be 50 or greater but there are exceptions)

Exclusion Criteria:

* Age less than 18 years old
* Patients unable to give informed consent
* Patients with history of colonic surgeries
* Patients with history of colonic motility disorder

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified by physicians in the endoscopy center at Vanderbilt. Those patients undergoing colonoscopy for either the indication of screening colonoscopy or IBD surveillance will be asked, on the day of their colonoscopy, whether they want to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yash Choksi, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center Endoscopy Laboratory, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Inflammatory Bowel Disease | Control
Started | 21 | 11
Completed | 21 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inflammatory Bowel Disease | Control | Total
Number analyzed (Participants) | 21 | 11 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 7 | 24
  >=65 years | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 18
  Male | 9 | 5 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 18 | 11 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 11 | 32

OUTCOME MEASURES:

1. Primary Outcome: Mucosal Impedance Values
Description: compare the mucosal impedance values between subjects with IBD and controls
Time Frame: 15 minutes
Population: Analysis is missing for 4 participants from each group either due to incomplete mucosal impedance (MI) readings or indeterminate disease status.
Measure: Median (Inter-Quartile Range); unit: ohms
Arm/Group | Inflammatory Bowel Disease | Control
Number analyzed (Participants) | 17 | 7
ohms
  Right Colon | 1139 [864 to 1347] | 849 [716 to 1250]
  Transverse Colon | 891 [705 to 1123] | 783 [752 to 880]
  Left Colon | 673 [547 to 763] | 699 [594 to 740]
  Rectum | 767 [618 to 991] | 531 [418 to 604]

2. Secondary Outcome: Difference in Inflamed and Normal Mucosa
Description: compare the mucosal impedance values in inflamed and normal areas in IBD patients
Time Frame: 15 minutes
Population: There were no patients where inflamed mucosa was directly adjacent to normal mucosa to be able to measure impedance in both
Arm/Group | Inflammatory Bowel Disease
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: After colonoscopy, patients are taken to the recovery area and monitored for complications as the sedative wears off. This time period is typically less than 60 minutes.
Arm/Group | Inflammatory Bowel Disease | Control
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/11
Other Adverse Events (participants affected / at risk) | 0/21 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-08): https://cdn.clinicaltrials.gov/large-docs/58/NCT03165058/Prot_SAP_000.pdf